CLINICAL TRIAL: NCT04661592
Title: Assessing Repeatability of the NeuroCatch Platform 2.0 Stimulus Sequences
Brief Title: NCP 2.0 Repeat Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCI_NCClin_004
Record Dates: First submitted 2020-11-17; First posted 2020-12-10 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Brain Health

STUDY DESIGN:
Intervention Model Description: Longitudinal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Experimental): Neurologically healthy individuals will be recruited for the longitudinal study
  Interventions: Device: NeuroCatch Platform

INTERVENTIONS:
Device: NeuroCatch Platform — To elicit the ERP components of interest in this study (N100, P300, N400), proprietary auditory stimulus sequences will be administered using the NeuroCatch™ Platform version 2.0, an investigational medical device. Each sequence consists of tones and word pairs to elicit the various components of interest. Version 2.0 of the NeuroCatch™ Platform consists of a computerized acquisition software which presents the stimulus, acquires the data and presents the amplitude and latency values of the ERP components (N100, N400, P300)

SUMMARY:
The NeuroCatch Platform™ version 2.0 (NCP2.0), an investigational medical device system developed by NeuroCatch Inc., consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP; brain response to a stimulus) information.

The purpose of the study is to understand how reliable and repeatable the ERP metrics elicited by the NCP platform are within participants over multiple sessions.

DETAILED DESCRIPTION:
A new method for creating stimulus sequences was developed for NeuroCatch™ Platform 2.0. Rather than using a set of fixed, predetermined sequences to elicit ERPs this new method draws on a database of candidate word stimuli to generate a different, random stimulus sequence each time a scan is carried out. The goal of this is to reduce habituation to the stimulus sequences which is hypothesized to improve the repeatability of the component measurements. Characterizing how individuals respond to the stimulus sequences is an important step in the validation of the generation method itself. Understanding the degree of variability and prototypical values of each ERP component is crucial to the understanding of typical brain functioning. For this type of technology to be clinically viable in quantifying brain health, the investigators must first quantify the degree to which a healthy brain naturally fluctuates in it processing capability. This study is being carried out to assess how repeatable the ERPs elicited by the new method are while also considering the impact of intraindividual variability observed in previous investigations. Thus, by comparing the results of the scans over time, an assessment of the reliability of the new stimulus sequences can be made.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex, at least 19 years of age or older
2. Able to understand the informed consent form, study procedures and willing to participate in study
3. Able to remain seated and focused for 7 minutes
4. In good health with no history of clinically relevant neurological illness or injury in the last 5 years

Exclusion Criteria:

1. Requires the use of hearing aids or a cochlear implant, diagnosed with tinnitus that is currently active, or has temporary damage to earing (e.g. punctured ear drum). Or unable to detect a 740Hz tone played at 85dB in both ears.
2. Implanted pacemaker or implanted electrical stimulators
3. Metal or plastic implants in the skull, excluding dental/facial implants
4. Exposed to an investigational drug or device 30 days prior to start in this study, or concurrent or planned use of investigational drug or device while enrolled in this study
5. Not proficient in English language
6. Diagnosed epilepsy or history of seizures
7. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
8. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in amplitudes of the N100 ERP acquired using the NeuroCatch™ Platform over 2 weeks - repeatability | Baseline, +1 Week, +2 Weeks
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the repeatability over three time points will be the intraclass correlation coefficient (ICC). Specifically, the two-way mixed single measures absolute agreement type of ICC (denoted as ICC(A,1)) will be used in this analysis.
Change in amplitudes of the N100 ERP acquired using the NeuroCatch™ Platform over 2 weeks - variability | Baseline, +1 Week, +2 Weeks
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the variability over three time points will be the group-mean of the individual standard deviations of the measures over the three time points
Change in Latency of the N100 ERP acquired using the NeuroCatch™ Platform over 2 weeks - repeatability | Baseline, +1 Week, +2 Weeks
  Latency (response speed) will be measured in milliseconds. The statistic being used to measure the repeatability over three time points will be the intraclass correlation coefficient (ICC). Specifically, the two-way mixed single measures absolute agreement type of ICC (denoted as ICC(A,1)) will be used in this analysis.
Change in Latency of the N100 ERP acquired using the NeuroCatch™ Platform over 2 weeks - variability | Baseline, +1 Week, +2 Weeks
  Latency (response speed) will be measured in milliseconds. The statistic being used to measure the variability over three time points will be the group-mean of the individual standard deviations of the measures over the three time points
Change in amplitudes of the P300 ERP acquired using the NeuroCatch™ Platform over 2 weeks - repeatability | Baseline, +1 Week, +2 Weeks
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the repeatability over three time points will be the intraclass correlation coefficient (ICC). Specifically, the two-way mixed single measures absolute agreement type of ICC (denoted as ICC(A,1)) will be used in this analysis.
Change in amplitudes of the P300 ERP acquired using the NeuroCatch™ Platform over 2 weeks - variability | Baseline, +1 Week, +2 Weeks
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the variability over three time points will be the group-mean of the individual standard deviations of the measures over the three time points
Change in Latency of the P300 ERP acquired using the NeuroCatch™ Platform over 2 weeks - repeatability | Baseline, +1 Week, +2 Weeks
  Latency (response speed) will be measured in milliseconds. The statistic being used to measure the repeatability over three time points will be the intraclass correlation coefficient (ICC). Specifically, the two-way mixed single measures absolute agreement type of ICC (denoted as ICC(A,1)) will be used in this analysis.
Change in Latency of the P300 ERP acquired using the NeuroCatch™ Platform over 2 weeks - variability | Baseline, +1 Week, +2 Weeks
  Latency (response speed) will be measured in milliseconds. The statistic being used to measure the variability over three time points will be the group-mean of the individual standard deviations of the measures over the three time points
Change in amplitudes of the N400 ERP acquired using the NeuroCatch™ Platform over 2 weeks - repeatability | Baseline, +1 Week, +2 Weeks
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the repeatability over three time points will be the intraclass correlation coefficient (ICC). Specifically, the two-way mixed single measures absolute agreement type of ICC (denoted as ICC(A,1)) will be used in this analysis.
Change in amplitudes of the N400 ERP acquired using the NeuroCatch™ Platform over 2 weeks - variability | Baseline, +1 Week, +2 Weeks
  Amplitude (response size) will be measured in microvolts. The statistic being used to measure the variability over three time points will be the group-mean of the individual standard deviations of the measures over the three time points
Change in Latency of the N400 ERP acquired using the NeuroCatch™ Platform over 2 weeks - repeatability | Baseline, +1 Week, +2 Weeks
  Latency (response speed) will be measured in milliseconds. The statistic being used to measure the repeatability over three time points will be the intraclass correlation coefficient (ICC). Specifically, the two-way mixed single measures absolute agreement type of ICC (denoted as ICC(A,1)) will be used in this analysis.
Change in Latency of the N400 ERP acquired using the NeuroCatch™ Platform over 2 weeks - variability | Baseline, +1 Week, +2 Weeks
  Latency (response speed) will be measured in milliseconds. The statistic being used to measure the variability over three time points will be the group-mean of the individual standard deviations of the measures over the three time points

SECONDARY OUTCOMES:
Collection and evaluation of adverse events and adverse device effects | At time of event
  Evaluation of safety and tolerability of the NeuroCatch™ Platform device
Change in hours of sleep of the day of scan | Baseline, +1 Week, +2 Weeks
  Secondary statistical analyses will explore the correlation between hours of sleep on the day of scan with changes in ERP measures (primary outcomes) across the sample
Change in perceived mood on the day of scan | Baseline, +1 Week, +2 Weeks
  Secondary statistical analyses will explore the correlation between perceived mood (ranked on a scale of 0-100) on the day of scan with changes in ERP measures (primary outcomes) across the sample

CONTACTS AND LOCATIONS:
Overall Officials: Jan Venter, MD, Principal Investigator — HealthTech Connex Inc.
Locations (1):
- HealthTech Connex Inc. Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No